CLINICAL TRIAL: NCT07188974
Title: Efficacy of Intra-Articular Injectable Platelet-Rich Fibrin (i-PRF) in the Treatment of Temporomandibular Joint Disorders
Brief Title: i-PRF for Temporomandibular Joint Disorders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Eskisehir Osmangazi University (Other)
Responsible Party: Principal Investigator, Gorkem Tekin, Asst.Prof., Eskisehir Osmangazi University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EskisehirOU-TEKIN-003
Record Dates: First submitted 2025-09-16; First posted 2025-09-23 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: TMJ Disc Disorder; Treatment; Arthrocentesis
Keywords: Injectable Platelet-Rich Fibrin (i-PRF); Pain Measurement; Mouth Opening
MeSH Terms: interventions — Arthrocentesis; proliferation regulatory factors, human urine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1: i-PRF Group (Experimental): Patients diagnosed with temporomandibular joint disorder will undergo arthrocentesis followed by intra-articular injection of i-PRF prepared from autologous blood.
  Interventions: Procedure: Arthrocentesis + Injectable Platelet-Rich Fibrin (i-PRF)
- Arm 2: Control Group (Active Comparator): Patients with temporomandibular joint disorder will undergo arthrocentesis only (joint lavage), without any additional intra-articular injection.
  Interventions: Procedure: Arthrocentesis (lavage only)

INTERVENTIONS:
Procedure: Arthrocentesis (lavage only) — A minimally invasive procedure in which the temporomandibular joint (TMJ) space is washed with sterile solution to remove inflammatory mediators and improve joint mobility.
  Arms: Arm 2: Control Group
Procedure: Arthrocentesis + Injectable Platelet-Rich Fibrin (i-PRF) — Autologous platelet-rich fibrin prepared by centrifugation of the patient's blood and injected intra-articularly into the TMJ following arthrocentesis. i-PRF contains platelets, leukocytes, and growth factors, which may promote tissue regeneration and healing.
  Arms: Arm 1: i-PRF Group

SUMMARY:
This study will evaluate whether intra-articular injectable platelet-rich fibrin (i-PRF) is more effective than arthrocentesis alone in treating temporomandibular joint (TMJ) disorders. Patients will be randomly assigned to two groups: one receiving arthrocentesis followed by i-PRF injection, and the other undergoing arthrocentesis only.

Pain intensity (VAS) and maximum mouth opening will be measured at baseline, 1 week, and 1 months. The goal is to determine if i-PRF provides greater pain relief and functional improvement compared with standard lavage.

DETAILED DESCRIPTION:
Temporomandibular joint (TMJ) disorders are a group of conditions that affect the jaw joint and surrounding muscles and ligaments. They can cause pain in the preauricular region, difficulty in opening or closing the mouth, clicking or crepitation sounds during movement, and impaired quality of life. Arthrocentesis, a minimally invasive procedure involving joint lavage, is often used when conservative treatments are not sufficient.

Injectable platelet-rich fibrin (i-PRF) is a second-generation platelet concentrate obtained from the patient's own blood without anticoagulants or additives. It contains high levels of platelets, leukocytes, and growth factors, which may promote tissue regeneration and healing. i-PRF has been used in various oral and maxillofacial procedures, and recent studies suggest that it may improve outcomes in TMJ disorders.

This randomized controlled trial aims to compare the effectiveness of intra-articular i-PRF injection with arthrocentesis alone in patients with TMJ disorders. Patients will be randomly assigned to one of two groups:

Experimental Group (i-PRF): Arthrocentesis followed by intra-articular injection of autologous i-PRF.

Control Group: Arthrocentesis only (joint lavage without any additional injection).

The primary outcome will be the change in pain intensity, measured using the Visual Analog Scale (VAS), and the secondary outcome will be the change in maximum mouth opening (measured in millimeters). Assessments will be performed at baseline, 1 week, and 1 months after treatment.

The study will be conducted at the Department of Oral and Maxillofacial Surgery, Eskişehir Osmangazi University, Turkey. It is expected that i-PRF will provide greater pain reduction and functional improvement compared to arthrocentesis alone, offering a regenerative and low-risk alternative in the management of TMJ disorders.

ELIGIBILITY:
Inclusion Criteria:

Patients ≥18 years old Diagnosed with temporomandibular joint disorder (TMD) based on clinical and radiological findings Presence of pain, restricted mouth opening, or joint sounds Voluntary participation and signed informed consent

Exclusion Criteria:

Systemic diseases affecting bone/joint healing (e.g., uncontrolled diabetes, rheumatoid arthritis, osteoporosis) Previous TMJ surgery or intra-articular injection Current pregnancy or breastfeeding Coagulopathy or anticoagulant therapy Allergy to hyaluronic acid (for control group) Inability to attend follow-up visits

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2024-09-02 (Actual); Primary Completion 2025-08-16 (Actual); Study Completion 2025-09-16 (Actual)

PRIMARY OUTCOMES:
Change in Pain Intensity (VAS score) | Baseline, 1 week, 1 month
  Pain intensity measured by Visual Analog Scale (VAS, 0-10).

SECONDARY OUTCOMES:
Change in Maximum Mouth Opening (mm) | Baseline, 1 week, 1 month
  Interincisal maximum mouth opening measured with a ruler in millimeters.

CONTACTS AND LOCATIONS:
Locations (1):
- Eskisehir Osmangazi University, Eskişehir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Comert Kilic S, Gungormus M. Is arthrocentesis plus platelet-rich plasma superior to arthrocentesis plus hyaluronic acid for the treatment of temporomandibular joint osteoarthritis: a randomized clinical trial. Int J Oral Maxillofac Surg. 2016 Dec;45(12):1538-1544. doi: 10.1016/j.ijom.2016.06.009. Epub 2016 Jun 28. PMID 27364372
- [Result] Moldez MA, Camones VR, Ramos GE, Padilla M, Enciso R. Effectiveness of Intra-Articular Injections of Sodium Hyaluronate or Corticosteroids for Intracapsular Temporomandibular Disorders: A Systematic Review and Meta-Analysis. J Oral Facial Pain Headache. 2018 Winter;32(1):53-66. doi: 10.11607/ofph.1783. Epub 2017 Dec 15. PMID 29244893